CLINICAL TRIAL: NCT02709993
Title: Phase I/II Study of Low-Dose Cyclophosphamide, Tumor Associated Peptide Antigen-Pulsed Dendritic Cell Therapy and Low Dose GM-CSF, As Consolidation Treatment in Patients With Hematologic Malignancies
Brief Title: Consolidation Therapy in Patients With Hematologic Malignancies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study unable to enroll patients
Sponsor: Kiromic BioPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KiroVAX001; BSK01 Dendritic cell vaccine (Other: Kiromic)
Record Dates: First submitted 2016-03-07; First posted 2016-03-16 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-08

CONDITIONS: Cancer; Hematologic Malignancies
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAPA-pulsed DC vaccine (Experimental): The subject will take low-dose cyclophosphamide by mouth for 5 days starting 7 days prior to the vaccine cycle. The vaccine contains 1 x 10^7 TAPA-pulsed dendritic cells and is administered SQ with low-dose GM-CSF following the low-dose cyclophosphamide cycle. A total of six (6) cycles of cyclophosphamide and six (6) DC vaccines cycles will be administered alternating every 14 days.
  Interventions: Biological: TAPA-pulsed DC vaccine

INTERVENTIONS:
Biological: TAPA-pulsed DC vaccine — A cycle of low-dose cyclophosphamide (100mg/day) by mouth for 5 days starting seven 7 days prior to the DC vaccine cycle to reduce Treg activity. Low-dose cyclophosphamide will be taken every 14 days for six 6 cycles. A total of 6 vaccines containing 1 x 10^7 TAPA-pulsed DC will be administered SQ every 14 days. The DC vaccine is given on Day 1 of the DCV cycle plus low-dose GM-CSF 50mcg/day SQ x 5 days (Day 1 to Day 4). GM-CSF is administered for 5 days to increase monocyte production and dendritic cell precursors to optimize immune responses.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Tumor Associated Peptide Antigen (TAPA) pulsed dendritic cell (DC) vaccines in the treatment of hematologic malignancies.

DETAILED DESCRIPTION:
Patients diagnosed with hematologic malignancies (as defined) who have responded to conventional therapy, and without any potentially curative therapeutic intervention, will be candidates for this Phase I/II study. Following confirmation of disease response to conventional antineoplastic therapy, eligible patients who agree to participate and sign a consent form will have their tumor cells and/or blood analyzed for the expression of a specific panel of Tumor Associated Peptide Antigens (TAPAs), including SP17, Ropporin, AKAP4, PTTG1 and Span-xb. Patients whose tumors express one (1) or more of these TAPAs will receive three (3) days of subcutaneous Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) to increase bone marrow production of monocytes and dendritic cell (DC) precursors, and peripheral blood mononuclear cells will be obtained by phlebotomy and/or leukapheresis for generation of autologous DCs. Patient's DCs will be generated at Kiromic's Cell Processing Good Manufacturing Process (GMP) facility, according to established Standard Operating Procedures, and activated by pulsing/loading them with the TAPA(s) relevant for each particular patient. Patients will receive five (5) days of low-dose cyclophosphamide prior to each vaccination with TAPA-pulsed DCs to decrease Treg activity. TAPA-pulsed DCs will be administered at a fixed dose of up to 1 x 107 DCs at least two (2) days following cyclophosphamide administration. DC vaccination schedule will be once every fourteen (14) days via subcutaneous (SC) and intradermal (ID) injections for a total of 6 vaccinations. Low dose GM-CSF will also be administered SC for five (5) consecutive days, starting three (3) to six (6) hours after each TAPA-pulsed DC treatment, to optimize immune response and DC viability in vivo. Patients will be followed on a weekly basis (or more frequently if required) to evaluate treatment-related toxicity. Immune responses and anti-tumor responses will be evaluated per protocol specifications. Continuation and stopping rules for the study will be defined based on toxicity/tolerability (Phase I) and/or immune responses (Phase II).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent.
2. Patients at least eighteen (18) years of age with histologically or cytologically proven Multiple Myeloma (MM), Hodgkins Disease (HD), Non-Hodgkins Lymphoma (NHL), Chronic Myelogenous Leukemia (CML), Acute Lymphocytic Leukemia (ALL), Acute Myelogenous Leukemia (AML) and Chronic Lymphocytic Leukemia (CLL), who have responded to standard, first-line antineoplastic therapy, as defined using standard response criteria for the specific hematologic malignancy (HM), and have no additional potentially curative therapeutic intervention available, will be eligible to participate in this study.
3. Expression of one (1) or more of the following TAPAs: SP17, AKAP4, Ropporin, PTTG1 and Span-xb, by either reverse transcriptase polymerase chain reaction (RT-PCR) and/or immunocytochemistry, Western blotting or ELISA, in neoplastic cells and/or blood.
4. Presence of measurable or evaluable disease (unless patient has achieved a complete response (CR) following first-line antineoplastic therapy).
5. Patients must not have any active infectious process.
6. Patients must have a negative test for HIV, Hepatitis A, B, and C.
7. Patients must not be receiving active immunosuppressive therapy.
8. Patients must have discontinued systemic antineoplastic therapy (including systemic corticosteroids and excluding tyrosine kinase inhibitors for CML) at least four (4) weeks prior to enrollment.
9. Patients may not have any known allergy to CYP and/or GM-CSF.
10. Patients must be willing to provide at least 250 mL, and up to 500 mL, of whole blood obtained by phlebotomy and/or consent to leukapheresis for DC generation.
11. Adequate renal and hepatic function (creatinine ≤ 2.0 mg/dl, bilirubin ≤ 2.0 mg/dl, aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 4X upper limit of normal range).
12. Adequate hematologic function (Platelets ≥ 60,000/mm3, lymphocytes ≥ 1,000/mm3, neutrophils ≥ 750/mm3, hemoglobin ≥ 10 g/dl).
13. Karnofsky performance status ≥ 70%.
14. Expected survival ≥ 6 months.
15. Patient Human Leukocyte Antigen (HLA) typing should demonstrate HLA-A*01, and/or HLA-A*02, and/or HLA-A*24 restriction.
16. Either a female or male of reproductive capacity wishing to participate in this study must be using, or agree to use, one or more types of birth control during the entire study and for 3 months after completing the study. Birth control methods may include condoms, diaphragms, birth control pills, spermicidal gels or foams, anti-gonadotropin injections, intrauterine devices (IUD), surgical sterilization, or subcutaneous implants. Another choice is for a subject's sexual partner to use one of these birth control methods. Women of reproductive capacity will be required to undergo a urine pregnancy test before completion of the post-screening informed consent process.

Exclusion Criteria:

1. Patients with HM, as previously defined, without confirmed response to standard, first-line antineoplastic therapy, and/or who do not fulfill all Inclusion Criteria as stated, will be ineligible to participate in this study.
2. Patients with HM who have undergone myeloablative systemic therapy are ineligible to participate in this study.
3. Patients without measurable or evaluable disease (unless patients achieved a complete response (CR) following 1st-line antineoplastic therapy).
4. Patients receiving cytotoxic therapy, radiation therapy, immunotherapy or non-topical steroids for HM within four (4) weeks of enrollment, excluding tyrosine kinase inhibitors in patients with CML.
5. Active immunosuppressive or cytotoxic therapy (excluding topical steroids) for any other condition.
6. Persistent fever (>24 hours) documented by repeated measurement or active, uncontrolled infection within 4 weeks of enrollment.
7. Active ischemic heart disease or history of myocardial infarction within six months.
8. Active autoimmune disease, including, but not limited to, Systemic Lupus Erythematosus (SLE), Multiple Sclerosis (MS), Ankylosing Spondylitis (AS), and Rheumatoid Arthritis (RA).
9. Pregnancy or breast feeding.
10. Patients with an active second invasive malignancy, other than basal cell carcinoma of the skin.
11. Life expectancy of less than 6 months.
12. Patients with contraindications to CYP and/or GM-CSF.
13. Patients who have received organ transplantations.
14. Patients with psychological or geographic conditions that prevent adequate follow-up or compliance with the study protocol.
15. Patients diagnosed with primary central nervous system (CNS) or with CNS metastases/involvement, at any time during the disease course, are excluded from the study.
16. Patients with HLA-A alleles not belonging to any of the following subtypes: HLA-A*01, or HLA-A*02, or HLA-A*24.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events due to administration of TAPA-pulse DC vaccine | every 7 days up to 5 months
  Number of adverse events due to administration of TAPA-pulse DC vaccine

SECONDARY OUTCOMES:
Immunological efficacy as indicated by T-cell cytokine levels | up to 5 months
  Immunological efficacy as indicated by T-cell cytokine levels
Immunological efficacy as determined by a positive delayed type hypersensitivity (DTH) skin test | up to 5 months
  Immunological efficacy as determined by a positive delayed type hypersensitivity (DTH) skin test

CONTACTS AND LOCATIONS:
Overall Officials: Naval G Daver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States